CLINICAL TRIAL: NCT04828928
Title: Prospective Study to Investigate Neuropathy in Patients Monitored for Wild-type TTR Cardiac Amyloidosis (Non-mutated)
Brief Title: Neuropathy in Patients Monitored for Wild-type TTR Cardiac Amyloidosis (Non-mutated)
Acronym: N-SAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/27
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Wild-type Amyloid Cardiopathy
Keywords: wild-type amyloid cardiopathy; neuropathy; descriptive study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- proportion of patients with neuropathy (Experimental): to prospectively study patients with a wild-type amyloid cardiopathy condition to identify and describe the associated neuropathy
  Interventions: Procedure: electromyogram

INTERVENTIONS:
Procedure: electromyogram — Patients meeting the criteria will be seen in consultation with standardized interview and clinical examination. An electromyogram will be then carried out to check for the presence of neuropathy. Finally, for patients diagnosed with neuropathy, a biological check-up to look for another cause of neuropathy will be performed. In patients who already had an EMG as part of their medical follow-up, the examination will not be repeated if it strictly meets the conditions of the minimum protocol and if it was done within the year prior to inclusion. In patients who already had an identical biological assessment in the year prior to inclusion, the sample will not be taken.

SUMMARY:
Transthyretin (TTR) amyloidosis is a rare disabling disorder that can be hereditary or sporadic. Depending on the form, various tissues are affected. While in hereditary cases, neuropathy is predominant, cardiac impairment is the main manifestation in the sporadic form.

The main objective of this project is to evaluate the proportion of patients with neuropathy in a population of patients with a non-mutated TTR amyloid cardiopathy condition.

DETAILED DESCRIPTION:
Transthyretin (TTR) amyloidosis belongs to a group of severe and multi-systemic diseases caused by an extracellular accumulation of fibrillar proteins arranged in beta-pleated sheets. This pathology can be hereditary (mutations in the TTR gene) or sporadic. Depending on the form, various tissues are affected: peripheral nervous system (leading to neuropathy, especially vegetative), heart, kidney... While in forms linked to TTR mutations neuropathy is the main manifestation, in the sporadic form (also called wild-type), the cardiac impairment is predominant. Other organ damages are rarely reported in this second form. In the THAOS registry (Coelho T. et al, 2013), a clinical peripheral neuropathy is reported in 28.4% out of 67 patients with the sporadic form of the disease, although the authors do not provide a precise description of the neuropathy type. We propose to prospectively study patients with a wild-type amyloid cardiopathy condition to identify and describe the associated neuropathy. A pilot study conducted at the Bordeaux University Hospital demonstrated the feasibility and interest of this research: it showed the presence of an undetermined aetiology polyneuropathy in 35.7% out of 14 patients followed for senile cardiac amyloidosis.

Tafamidis is used on familial amyloid neuropathy and a recent study shows an effect on senile amyloid cardiopathy (Maurer MS et al., 2018) which strengthens the need to determine the frequency of neuropathies associated with wild-type amyloid cardiopathy and to type them more accurately.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both gender, over 18 years old, with transthyretin amyloid cardiopathy according to one of the two American Heart Association definitions of 2016
* No mutation in the TTR gene
* Patients giving their free and informed consent to participate after information about the research
* Patients affiliated to or benefiting from a social security scheme

Exclusion Criteria:

* Patients with chronic neuropathy related to a known aetiology
* Patients under guardianship or curatorship

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Presence of a clinical and/or electrophysiological neuropathy | within 6 months of inclusion (at the time of the electromyogram)
  The diagnosis of peripheral neuropathy should meet P.J. Dyck's definition of peripheral neuropathy (New England Journal of Medicine, 1982), based on:
  * the clinical judgment resulting from the standardized clinical examination (carried out by an expert neurologist) and according to the HAS recommendations on the diagnosis of peripheral neuropathies;
  * electrophysiological abnormalities, interpreted in the clinical context, after an examination carried out by an expert neurophysiologist.

SECONDARY OUTCOMES:
Clinical data of patients with polyneuropathy with no identified etiology: Epidemiological characteristics | within 6 months of inclusion (at the time of the electromyogram)
  age, sex, age at diagnosis, age at assessment
Clinical data of patients with polyneuropathy with no identified etiology: history characteristics | within 6 months of inclusion (at the time of the electromyogram)
  carpal tunnel, diabetes, narrow cervical canal, alcohol consumption, radiculalgia in the lower limbs
Clinical data of patients with polyneuropathy with no identified etiology: Heart attack | within 6 months of inclusion (at the time of the electromyogram)
  Heart failure ( yes/no), pacemaker (Yes/no) and Functional classification of heart disease according to the New York Heart Association (NYHA) score.
  The NYHA score is a classification in 4 stages of increasing severity is proposed by the New York Heart Association, it is based on the intensity of the symptoms:
  I: Asymptomatic, discomfort during exceptional efforts. II: Moderate discomfort for significant efforts. III: Discomfort felt during moderate efforts. IV: Discomfort during the slightest effort or at rest. Référence: Hurst Hurst JW, Morris DC, Alexander RW. The use of the New York Heart Association's classification of cardiovascular disease as part of the patient's complete Problem List. Clin Cardiol . JW, Morris DC, Alexander RW. L'utilisation de la New York Heart Association de classification du des maladies cardiovasculaires dans le cadre du patient compléter la liste des problèmes. Clin Cardiol. 1999 Jun ;22 (6):385-90.
Clinical data of patients with polyneuropathy with no identified etiology: Clinical scores - KARNOFSKI index | within 6 months of inclusion (at the time of the electromyogram)
  The KARNOFSKY index is used to assess the general condition of the patient: it is a scale from 0 to 100, the maximum representing the absence of complaints related to the disease.
Clinical data of patients with polyneuropathy with no identified etiology: Clinical scores - NIS-LL- | within 6 months of inclusion (at the time of the electromyogram)
  Neuropathy Impairment Score-Lower Limb (NIS-LL): this is a score out of 88, the minimum (0) representing an asymptomatic patient
Clinical data of patients with polyneuropathy with no identified etiology: Clinical scores - ONLS- | within 6 months of inclusion (at the time of the electromyogram)
  The Overall Neuropathy Limitation Scale (ONLS) is used to assess the functional impact of neuropathy: score out of 12, the minimum (0) representing a patient without any functional impairment related to his neuropathy.
Clinical data of patients with polyneuropathy with no identified etiology: Clinical scores - RODS- | within 6 months of inclusion (at the time of the electromyogram)
  The Rasch Score-built Overall Disability Scale (RODS) is used to assess the impact of neuropathy on activities of daily living: it is a scale from 0 to 48 with the maximum representing a patient asymptomatic.
Clinical data of patients with polyneuropathy with no identified etiology: Clinical scores - CADT- | within 6 months of inclusion (at the time of the electromyogram)
  The Compound Autonomic Dysfunction Test (CADT) is used to assess vegetative impairment: it is rated out of 16 maximum if normal (erectile dysfunction will not be taken into account in men).
Clinical data of patients with polyneuropathy with no identified etiology: Clinical scores -MoCA- | within 6 months of inclusion (at the time of the electromyogram)
  The Montreal Cognitive Assessment (MoCA) is used for a cognitive assessment: out of 30, the maximum being a subject without impairment.
Clinical data of patients with polyneuropathy with no identified etiology: Electrophysiological data | within 6 months of inclusion (at the time of the electromyogram)
  This data includes:
  * Motor and / or sensory impairment
  * Axonal and / or demyelinating character
  * Length-dependent or non-length-dependent character
  * Topography of the disease
Estimation of the frequency of the presence of neuropathy in our study population in order to compare it to a reference population | 24 months
  Estimation of the frequency of the presence of neuropathy in our study population in order to compare it to a reference population

CONTACTS AND LOCATIONS:
Overall Officials: Guilhem SOLE, MD, Principal Investigator — Université Hospital, Bordeaux
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHU de Nantes, Nantes
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No